CLINICAL TRIAL: NCT00145223
Title: Research for Elimination of Human Filariasis
Brief Title: Research for Elim of Filariasis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 00-015
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: W. Bancrofti Filariasis
Keywords: Wuchereria bancrofti, filariasis, Egypt
MeSH Terms: conditions — Filariasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Wuchereria bancrofti, is a mosquito-transmitted parasite that causes deforming lymphatic filariasis in the tropics. Improved treatment methods have led to new thinking that it should be possible to interrupt transmission and eliminate this major public health problem by repeated, annual cycles of mass treatment with new single dose combination drug regimens. Egyptian villages involved in the study will be surveyed. Household members above 4 years of age will be tested for filariasis. Also, children in the first year classes of primary schools (5 to 6 years of age) will be tested for parasite infection. Village populations will be treated for filariasis as part of the MOH national filariasis elimination program. Children under age 5, pregnant women, and people with severe underlying illness are excluded from the program.

DETAILED DESCRIPTION:
Approximately 100 million people are infected with Wuchereria bancrofti, a mosquito-transmitted nemotade parasite that causes deforming lymphatic filariasis in the tropics. Improved therapies and diagnostic methods have led to new thinking about lymphatic filariasis and the realization that it should be possible to interrupt transmission and eliminate the major public health problem by repeated, annual cycles of mass treatment with new single dose combination drug regimens. The Egyptian Ministry of Health is about to institute annual mass therapy with Albendazole (ALB) and diethylcarbamazine (DEC) in all filariasis endemic villages in the country with the aim of eliminating filariasis. This study comprises 4 different activities involving human subjects: These are Village studies of filariasis prevalence and intensity, school studies of antibody prevalence, A treatment trial with an assessment of infectivity of humans with mosquito feeding before and after treatment. Pre-control evaluations of villages will be performed in year 1. Mass treatment will be conducted annually by the MOH, beginning late in year one or early in year 2. Timing of annual follow-up evaluations in years 2-4 will be coordinated with the MOH so that specimens are collected at least 6 months after mass treatment but prior to the next distribution of medication. It is anticipated that the third follow-up collection will be completed by the end of year 4. A final set of follow-up specimens will be collected in year 5 if time permits. The treatment trial will compare effects of diethylcarbamzine (6 mg/kg) and albendazole (400 mg) given as a single dose, 7 consecutive daily doses, or once weekly for 4 weeks. Antibody prevalence in young children (school studies), 200-300/school; infection prevalence studies (village studies sampling humans and mosquitoes), 100 houses (approx. 500 people) per village; treatment trial, n = 60 (20 per treatment group). The project will attempt to measure effects of mass therapy with tools developed in prior studies. It is anticipated that infection prevalence rates and infection intensities will decrease following mass therapy. A successful program should lead to elimination of filariasis over time.

ELIGIBILITY:
Inclusion Criteria:

For village prevalence studies, subjects must reside in villages that are endemic for lymphatic filariasis with MF prevalence rates greater than or equal to 5%. For school studies, subjects must live in endemic villages and attend primary schools.

Exclusion Criteria:

Village studies: Age less than 5 years. School studies: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-08; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt